CLINICAL TRIAL: NCT01924169
Title: A Study of Immune-adjuvant Effect of Lenalidomide in Patients With Chronic Lymphocytic Leukemia and Hypogammaglobulinemia and Impaired Response to Vaccinations - RV-CL-CLL-PI-002544
Brief Title: Lenalidomide as Immune Adjuvant in Patient's With Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-0371; NCI-2014-01058 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Hematologic Disorder
Keywords: Hematologic Disorder; Chronic Lymphocytic Leukemia; CLL; Hypogammaglobulinemia; Impaired Response to Vaccinations; Immunoglobulins; Immune system's function; Lenalidomide; CC-5013; Revlimid; Flu vaccine; TIV; Pneumonia vaccine
MeSH Terms: conditions — Hematologic Diseases; Leukemia, Lymphocytic, Chronic, B-Cell; Agammaglobulinemia; Influenza, Human | interventions — Lenalidomide; Influenza Vaccines; SARS-CoV-2 inactivated vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide administered at the dose of 5 mg/day on Monday, Wednesday and Friday for 3 months. If Immunoglobulin G (IgG) levels improve by at least 25% of baseline, lenalidomide administration continued for 3 months on, and 3 months off for 2 years. If IgG levels do not improve, frequency of lenalidomide increased to 5 mg/day for additional 3 months and if response is achieved, lenalidomide continued at 5mg/day 3 month on/3 month off for a total of 2 years. Seasonal influenza vaccination (Trivalent Influenza Vaccine, Fluzone High Dose) administered yearly, during the fall/winter season and pneumococcal immunization (Pneumococcal Polysaccharide Vaccine, Pneumovax) administered once between month 6 and month 21.
  Interventions: Drug: Lenalidomide; Biological: Influenza Vaccine; Biological: Pneumovax Vaccine

INTERVENTIONS:
Drug: Lenalidomide — 5 mg/day by mouth on Monday, Wednesday and Friday for 3 months. Process repeated for up to 2 years.
  If IgG levels do not improve, frequency of lenalidomide increased to 5 mg/day by mouth for additional 3 months and if response is achieved, lenalidomide continued at 5mg/day 3 month on/3 month off for a total of 2 years.
  Other Names: CC-5013; Revlimid
Biological: Influenza Vaccine — Administered as injection yearly, during the fall/winter season.
  Other Names: TIV
Biological: Pneumovax Vaccine — Administered by injection once between month 6 and month 21. Patients, who have received the Pneumovax vaccine within last 5 years, will not receive Pneumovax vaccination.
  Other Names: Pneumonia vaccine

SUMMARY:
The goal of this clinical research study is to learn if lenalidomide can increase the level of immunoglobulins (parts of the blood that may help to improve the immune system's function) and/or will improve the protective effect of the flu and pneumonia vaccines in patients with CLL.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take lenalidomide by mouth on Monday, Wednesday and Friday for 3 months.

In order to participate in this study you must register into and follow the requirements of the Revlimid REMS™ program of Celgene Corporation. This program provides education and counseling on the risks of fetal exposure, blood clots and reduced blood counts. You will be required to receive counseling every 28 days during treatment with lenalidomide, follow the pregnancy testing and birth control requirements of the program that are appropriate for you and take telephone surveys regarding your compliance with the program.

Depending on how you respond to the drug, after 3 months, you will either:

°Take lenalidomide every Monday, Wednesday and Friday on a 3 months on/3 months off schedule. You will then repeat this process for up to 2 years.

or

°Take lenalidomide every day for an extra 3 months. If you respond well, you will take lenalidomide every day for 3 months, then for the next 3 months stop the drug. You will then repeat this process for up to 2 years.

You should swallow the lenalidomide capsules whole with water. Do not open, crush, or break the lenalidomide capsules. If you touch a broken lenalidomide capsule, wash the area of your body with soap and water.

If you miss a dose of lenalidomide, and it has been less than 12 hours since your regular dose time, take it as soon as you remember. If it has been more than 12 hours, just skip your missed dose. Do not take 2 doses at the same time. If you take too much lenalidomide or overdose, call your healthcare provider right away. If you vomit after any dose, do not take another dose.

You will also receive a vaccine for the flu (Trivalent or Fluzone) 1 time a year. If you have not received one in the last 5 years, you will receive a vaccine for pneumonia (Pneumovax) between months 6 and 21. You will receive these vaccines as an injection under the skin.

Study Visits:

Before the first dose of study drug:

°Blood (about 2 teaspoons) will be drawn to test cytokines (proteins that may affect the immune system) and to test your immune system.

If you are able to become pregnant, 1 time a week for the first 4 weeks and then every 28 days while on treatment, you will have a blood (about 1 teaspoon) or urine pregnancy test.

While you are taking lenalidomide, blood (about 1 teaspoon) will be drawn for routine tests every 2-4 weeks.

At 3 months (+/- 3 weeks):

* You will have a physical exam.
* Blood (about 1 teaspoon) will be drawn for routine tests.

Before the flu vaccine, blood (about 1 teaspoons) will be drawn for antibody testing. Antibodies are created by the immune system and may attack foreign cells or substances, such as the study drug.

At 4 weeks (+/- 2 weeks) and 3 months (+/- 3 weeks) after the vaccine, blood (about 2 teaspoons) will be drawn for antibody testing, cytokine testing, and to test your immune system.

Length of Study:

You will take the study drug for up to 2 years. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End of Study:

°Blood (about 2 teaspoons) will be drawn for antibody testing and cytokine testing.

This is an investigational study. Lenalidomide is FDA approved and commercially available for the treatment of multiple myeloma, myelodysplastic syndrome and mantle cell lymphoma. The use of this to help prevent infections by improving immunoglobulin levels and its use in combination with the flu and pneumonia vaccine is investigational.

Up to 35 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic lymphocytic leukemia (CLL) patients with IgG less than 500 mg/dl with/without symptoms who are either untreated or previously treated, regardless of response, at least 6 months from prior therapy (including mAb)..
2. Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status of 0-2.
3. Adequate renal functions as indicated by serum creatinine equal to or less than 2 mg/dl.
4. Adequate hepatic function indicated as total bilirubin equal to or less than 2 mg/dl and alanine aminotransferase (ALT) equal to or less than two times the upper limit of normal.
5. Disease free of prior malignancies for 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. Patients with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery can be enrolled in the study as long as they have a reasonable expectation to have been cured with the treatment modality received.
6. Females of childbearing potential (FCBP). A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has not had menses at any time in preceding 24 consecutive months)>
7. FCBP must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mlU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide.
8. FCBP must also agree to ongoing pregnancy testing (weekly for the first four weeks and then every 28 days while on therapy and at discontinuation of treatment).
9. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
10. Patients must be 18 years of age or older.
11. All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
12. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

1. Known sensitivity to lenalidomide or other thalidomide derivatives.
2. History of Guillain-Barre within 6 weeks of previous influenza vaccination.
3. Patient on steroid therapy.
4. Documented prolymphocytic leukemia (prolymphocytes more than 55% in the blood) or Richter's transformation.
5. Known positivity for HIV or active hepatitis B or C.
6. Pregnant or breast feeding females.
7. History of tuberculosis treated within the last five years or recent exposure to tuberculosis.
8. Any serious medical condition, laboratory abnormality or psychiatric illness that places the subject at unacceptable risk if he/she were to participate in the study.
9. Patients with a recent history of deep vein thrombosis (DVT) or pulmonary embolus (PE), in six months prior to enrollment are not eligible for this study.
10. Subjects who have currently active hepatic or biliary disease (with the exception of patients with Gilbert's syndrome).
11. Patients with severe allergic reaction (e.g., anaphylaxis) after previous dose of any influenza vaccine or to a vaccine component, including egg protein.
12. Moderate or severe acute illness with or without fever.
13. Use of any other experimental drug or therapy within 28 days of baseline.
14. Concurrent use of other anti-cancer agents or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD,BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 2014 through May 2016. All of the participants were recruited at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Lenalidomide: Lenalidomide administered at the dose of 5 mg/day three times a day for three months. If IgG levels improve by at least 25% of baseline, lenalidomide administration continued for 3 months on, and 3 months off for 2 years. If Immunoglobulin G (IgG) levels do not improve, frequency of lenalidomide increased to 5 mg/day for additional 3 months and if response is achieved, lenalidomide continued at 5mg/day 3 month on/3 month off for a total of 2 years.
  Seasonal influenza vaccination (Trivalent Influenza Vaccine, Fluzone High Dose) administered yearly, during the fall/winter season and pneumococcal immunization (Pneumococcal Polysaccharide Vaccine, Pneumovax) administered once between month 6 and month 21.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Lenalidomide: Lenalidomide administered at the dose of 5 mg/day three times a day for three months. If IgG levels improve by at least 25% of baseline, lenalidomide administration continued for 3 months on, and 3 months off for 2 years. If IgG levels do not improve, frequency of lenalidomide increased to 5 mg/day for additional 3 months and if response is achieved, lenalidomide continued at 5mg/day 3 month on/3 month off for a total of 2 years.
  Seasonal influenza vaccination (Trivalent Influenza Vaccine, Fluzone High Dose) administered yearly, during the fall/winter season and pneumococcal immunization (Pneumococcal Polysaccharide Vaccine, Pneumovax) administered once between month 6 and month 21.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 65 [48 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With IgG Response
Description: IgG response defined as having improvement in IgG level by at least 25% at 6 months, compared to baseline.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Seroconversion Response
Description: Study considered positive in regard to the secondary endpoints if seroconversion is observed in 60% or more of the subjects for at least one of the vaccinations given.
Time Frame: 4 weeks after flu vaccine administered
Population: The first three participants did not remain on study long enough to undergo immunizations.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants will be assessed for adverse events from the first dose of study medication to the completion of study treatment, up to 6 months.
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=3)
Fatigue/Malaise (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
insomnia (Nervous system disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-07-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT01924169/Prot_000.pdf
  • Statistical Analysis Plan (2013-07-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT01924169/SAP_001.pdf